CLINICAL TRIAL: NCT02035631
Title: Prevention of Breast Cancer Recurrence Through Weight Control, Diet, and Physical Activity Intervention
Acronym: PREDICOP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREDICOP
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Breast Neoplasms; Recurrence
Keywords: Breast Neoplasms; Recurrence; Motor Activity; Diet; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Recurrence; Motor Activity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Lifestyle intervention combining weight control, diet and physical activity
  Interventions: Behavioral: Diet; Behavioral: Physical activity
- Minimal intervention (Sham Comparator): Minimal diet intervention and minimal physical activity intervention
  Interventions: Behavioral: Minimal diet intervention; Behavioral: Minimal physical activity intervention

INTERVENTIONS:
Behavioral: Diet — The dietary component, aimed to reduce calorie intake according to individual requirements, will be structured in 1-hour weekly sessions led by trained nutritionists. Sessions will concentrate on teaching participants about food groups, the food pyramid and Mediterranean diet, how to chose, prepare and cook hypo-caloric meals.
  Arms: Intervention
Behavioral: Physical activity — The physical activity component will include two sessions per week led by trained physical activity monitors including aerobic exercise of high/moderate intensity, and instruction about the at-home exercise activities (3 more sessions).
  Arms: Intervention
Behavioral: Minimal diet intervention — Some basic diet recommendations
  Arms: Minimal intervention
Behavioral: Minimal physical activity intervention — Some basic recommendations on physical activity
  Arms: Minimal intervention

SUMMARY:
The main purpose of our study is to assess the effect of a lifestyle intervention combining weight control, diet and physical activity on the risk of recurrences among breast cancer patients with non-metastatic tumours in terms of 5-year cumulative incidence of recurences.

DETAILED DESCRIPTION:
BACKGROUND/MAIN OBJECTIVE: The main purpose of our study is to assess the effect of a lifestyle intervention combining weight control, diet and physical activity on the risk of recurrences among breast cancer patients with non-metastatic tumours. As secondary objectives we aim to assess whether the proposed intervention is able to improve the overall survival or the disease-free survival, as well as quality of life of breast cancer patients. METHODOLOGY: This multicentric randomized controlled trial aims to include 2108 women (1054 per arm), aged up to 75 years, diagnosed with a non-metastatic breast cancer (stage I, II, IIIA) in the participating centres, whose standard treatment was completed within the last 3 months. Participants will be assigned to either an intervention or a control group, and followed for five years. Patients assigned to the control arm will continue with the usual care, including standard guidelines for weight control applied in the centre. Patients in the intervention group will be involved in a lifestyle program with two components. The dietary part will aim to achieve a calorie reduction while maintaining nutritional quality; the physical activity part will include supervised sessions of moderate intensity. Data will be analyzed on an intention to treat basis using time-toevent analysis. HYPOTHESES: We expect a significant reduction in the 5-year cumulative incidence of recurrences (primary outcome) in the intervention group. Furthermore, as secondary outcomes, we expect a significant increase in overall survival and an improvement of quality of life of patients included in the intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* incident primary breast cancer (ICD-O C50)
* stage at diagnosis I, II, IIIA (or T1-3, N0-N2, M0)
* age at diagnosis below 76 years
* within 3 months since completion of standard treatment (excluding hormonal therapy) and within 15 months since the diagnosis of the disease

Exclusion Criteria:

* morbid obesity (BMI >40kg/m²) or underweight (BMI <18kg/m²)
* ischemic heart disease (coronary syndrome, unstable angina or myocardial infarction) or cerebrovascular incident (ischemic or hemorrhagic) during the previous 12 months
* diabetes (only if unstable - glycosylated haemoglobin >9%)
* current medical or surgical treatment to lose weight
* mental illness that would prevent the patient from carrying out the intervention
* logistical factors which would prevent the patient from carrying out the intervention (distance to travel, work or family commitments)
* pregnant or planning pregnancy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2014-01; Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Time to local and distant recurrence | 5 years from recruitment day
  Time between recruitment date and local and distant recurrence date or end of the 5-year follow-up which ever occurs first

SECONDARY OUTCOMES:
Overall survival | 5 years
  Time between recruitment date and death date or end of 5-year follow-up which ever occurs first
Disease free survival | 5 years
  Time between recruitment date and recurrence (local or distant) or death or end of 5-year follow-up which ever occurs first
Quality of life | Baseline, one year and three years
  Quality of life assessments using the SF36, the FACIT (fatigue questionnaire) and the HADS (Anxiety and depression)

OTHER OUTCOMES:
Changes in biomarkers | Baseline and one year
  Biomarkers related to:
  * sex hormone profile,
  * dietary intake,
  * insulin resistance,
  * inflammation process
  * and any biomarker possibly related to the progression of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Cirauqui Cirauqui, MD, Principal Investigator — Fundació Institut d'Investigació Germans Trias i Pujol; Sonia Del Barco Berron, MD, Principal Investigator — Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta; Vanesa Ortega Cebrián, MD, Principal Investigator — Hospital Vall d'Hebron; Maria Angeles Arcusa Lanza, MD, Principal Investigator — Consorci Sanitari de Terrassa; Antonio Agudo, MD, Principal Investigator — Institut Català d'Oncología - L'Hospitalet (ICO)
Locations (5):
- Spain (5):
  - Fundació Institut d'Investigació Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Institut Catala d'Oncologia - L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta, Girona, Girona